CLINICAL TRIAL: NCT05220397
Title: A Phase III, Prospective, Open-Label, Randomized Clinical Trial Evaluating the Augmenting of Anti-SARS-CoV2 Immunity in Kidney Transplant Recipients Via a Heterologous Additional Dose With Janssen Ad26.CoV2.S Vaccine
Brief Title: Janssen Ad26.CoV2.S Vaccine Booster in Kidney Transplant Recipients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Janssen Biotech, Inc stopped production of the vaccine, and it was no longer available as of 2023.
Sponsor: Mark Stegall (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor-Investigator, Mark Stegall, Sponsor-Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 21-008036
Record Dates: First submitted 2022-01-27; First posted 2022-02-02 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Kidney Transplant Recipient
Keywords: kidney transplant; renal transplant; COVID-19; COVID-19 vaccine; Janssen Ad26.CoV2.S vaccine; adenovector vaccine
MeSH Terms: conditions — COVID-19 | interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Initial Responders (No Intervention): Individuals who have previously received the Pfizer or Moderna vaccines and have high levels of spike antibodies in their blood, will receive standard of care immunosuppressive (IS) medications.
- Low Level (LL) Spike Antibodies: Janssen Vaccine Responders (Experimental): Individuals who had a spike protein test result less than 250 U/mL at the screening visit. Subjects received one dose of the Janssen Ad26.CoV2.S vaccine. After receiving the Janssen Ad26.CoV2.S vaccine, their spike protein test results were greater than or equal to 250 U/mL.
  Janssen Ad26.CoV2.S Vaccine: Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
  Interventions: Biological: Janssen Ad26.CoV2.S Vaccine
- Low Level (LL) Spike Antibodies: Janssen Vaccine Non-Responders (Experimental): Individuals who had a spike protein test result less than 250 U/mL at the screening visit. Subjects received one dose of the Janssen Ad26.CoV2.S vaccine. After receiving the Janssen Ad26.CoV2.S vaccine, their spike protein test results were less than 250 U/mL. 28 days following the first dose of the Janssen Ad26.CoV2.S vaccine, subjects were given a second dose of Janssen Ad26.CoV2.S vaccine.
  Janssen Ad26.CoV2.S Vaccine: Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
  Interventions: Biological: Janssen Ad26.CoV2.S Vaccine
- Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication (Experimental): Individuals who had a spike protein test result less than 250 U/mL at the screening visit. Subjects were randomized to maintain their current immunosuppression medication regimen and then receive a Janssen Ad26.CoV2.S vaccine. 28 days after receiving the first dose of the Janssen Ad26.CoV2.S vaccine, if a subject's spike protein test results were less than 250 U/mL then a second dose of the Janssen Ad26.CoV2.S vaccine was administered.
  Janssen Ad26.CoV2.S Vaccine: Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
  Maintenance in Immunosuppression Medication: Maintain current immunosuppression medication dosage
  Interventions: Biological: Janssen Ad26.CoV2.S Vaccine; Other: Maintenance in Immunosuppression Medication
- Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication (Experimental): Individuals who had a spike protein test result less than 250 U/mL at the screening visit. Subjects were randomized to change their current immunosuppression medication regimen and then receive an additional Janssen Ad26.CoV2.S vaccine.
  Janssen Ad26.CoV2.S Vaccine: Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
  Reduction in Immunosuppression Medication: Reduction in immunosuppression medication dosage
  Interventions: Biological: Janssen Ad26.CoV2.S Vaccine; Other: Reduction in Immunosuppression Medication

INTERVENTIONS:
Biological: Janssen Ad26.CoV2.S Vaccine — Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
  Arms: Low Level (LL) Spike Antibodies: Janssen Vaccine Non-Responders; Low Level (LL) Spike Antibodies: Janssen Vaccine Responders; Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication; Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication
Other: Reduction in Immunosuppression Medication — Reduction in immunosuppression medication dosage
  Arms: Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Other: Maintenance in Immunosuppression Medication — Maintain current immunosuppression medication dosage
  Arms: Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication

SUMMARY:
The purpose of this research is to see if a dose of the Janssen Ad26.CoV2.S vaccine effects the immune protection in individuals who have had a kidney transplant and two or three doses of mRNA vaccine (Pfizer and/or Moderna vaccines).

DETAILED DESCRIPTION:
Early after receiving an messenger ribonucleic acid (mRNA) COVID-19 vaccination, most of the general population achieves an anti-COVID spike protein antibody >250 U/ml. A large percentage of transplant patients form no anti-COVID spike protein antibody or have levels <250U/ml even early after vaccination. While a direct correlation between any specific anti-COVID spike protein antibody has not been studied extensively, transplant patients do appear to have higher rates of COVID infections and possibly higher mortality rates.

Thus, 250 U/ml (the saturation level of the assay below which does not require dilutions) is the target level of anti-COVID spike protein antibody, as that will be considered a "normal" response to the vaccine in this clinical trial. There is no data for intermediate levels of antibody (likely the higher the better the protection). In the absence of any intermediate level data, this study aims to achieve a normal response in transplant recipients receiving the Janssen Ad26.COV2.S vaccine.

This study is a phase III, prospective, open label clinical trial with one randomized arm. Its goal is to meet the unmet clinical need to provide vaccine induced immunity for immunocompromised kidney transplant patients after receiving two or three doses of the Pfizer or Moderna COVID-19 vaccine.

ELIGIBILITY:
Inclusion Criteria:

Criteria for Entry into the Study:

* Any kidney transplant recipient from Mayo Clinic who has received the mRNA vaccine (two or three dose mRNA vaccine-Moderna or Pfizer) and are >28 days after most recent vaccination at the time of spike protein assessment.
* Recipients of a kidney transplant, including those transplanted with other solid organ transplants in addition to the kidney. Subjects may have received more than 1 kidney transplant.
* More than 90 days since any transplant including a kidney transplantation. •≥18 years of age on the day of consent.

Criteria for Entry into Segment I

* Must have a Roche Elecsys® Anti-SARS-CoV-2 S level of <250 U/mL to be eligible for Segment I.
* Platelet count of >75,000/µL on the day of vaccination with the Janssen Ad26.CoV2.S vaccine.
* Contraceptive (birth control) use should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies.
* Before randomization, participants must be either:

  * Not be of childbearing potential
  * Of childbearing potential and practicing an acceptable effective method of contraception. Subject must agree to remain on contraception from date of consent until 3 months after the last dose of the Janssen Ad26.CoV2.S vaccine. Use of hormonal contraception should start at least 28 days before the 1st administration of the Janssen Ad26.CoV2.S vaccine. The sponsor-investigator should evaluate the potential for contraceptive method failure (for example, noncompliance, recently initiated) in relationship to the Janssen vaccination. Acceptable effective method for this study include:

    * Hormonal contraception:

      * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
      * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
    * Intrauterine device
    * Intrauterine hormone-releasing system
    * Bilateral tubal occlusion/ligation procedure
    * Vasectomized partner (the vasectomized partner should be the sole partner for that participant)
    * Sexual abstinence (defined as refraining from heterosexual intercourse from the date of consent until 3 months after the last dose of the Janssen Ad26.CoV2.S vaccine. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant.). Note: Use of condoms is not considered as an acceptable contraceptive barrier method due to the failure rate of female and male condoms (Centers for Disease Control and Prevention. Reproductive Health: Contraception. https://www.cdc.gov/reproductivehealth/contraception/index.htm. Accessed 23 November 2020)
* If subject is female and of childbearing potential, she must:

  * Have a negative highly sensitive serum pregnancy test prior to vaccination.
* Participant agrees to not donate bone marrow, blood, and blood products from the first Janssen Ad26.CoV2.S vaccine administration until 3 months after the last dose of the Janssen Ad26.CoV2.S vaccine.

Exclusion Criteria:

* Clinically significant acute illness (this does not include minor illnesses such as diarrhea or mild upper respiratory tract infection) or temperature ≥38.0ºCelsius (C) (100.4°Fahrenheit [F]) within 24 hours prior to the planned 1st dose of the Janssen Ad26.CoV2.S vaccine; randomization at a later date is permitted at the discretion of the sponsor-investigator.
* Has a known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the Janssen Ad26.CoV2.S vaccine; refer to the Investigative Brochure).
* Subject has received or plans to receive:

  * Licensed live attenuated vaccines -within 28 days before or after planned administration of the 1st or subsequent Janssen vaccinations.
  * Other licensed (not live) vaccines -within 14 days before or after planned administration of the 1st or subsequent Janssen vaccinations.
* Received an investigational drug within 30 days (including investigational drugs for prophylaxis of COVID-19) or used an invasive investigational medical device within 30 days of the Janssen Ad26.CoV2.S vaccine. Received investigational Ig or investigational monoclonal antibodies within 3 months, or received convalescent serum for COVID-19 treatment within 4 months or received an investigational vaccine (including investigational Adenoviral- vectored vaccines) within 6 months before the planned administration of the 1st dose of the Janssen Ad26.CoV2.S vaccine or is currently enrolled or plans to participate in another investigational study within 3 months after the last Jansen vaccination.

Note: Participation in an observational clinical study is allowed at the sponsor-investigator's discretion; please notify the sponsor-investigator of this decision. Efforts will be made to ensure inclusion of participants who have not been previously enrolled in coronavirus studies. In order to participate subject must agree and understand that they cannot enroll in other coronavirus focused studies while participating in this one.

* Is pregnant or planning to become pregnant at the time of consent and within 3 months of the last dose of the Janssen Ad26.CoV2.S vaccine.
* Has a history of an underlying clinically significant acute or chronic medical condition or physical examination findings which, in the opinion of the sponsor-investigator, would make study participation not be in the participant's best interest (e.g., compromise the well- being) or that could prevent, limit, or confound the protocol-specified assessments.
* Has a contraindication to Intramuscular (IM) injections and blood draws.
* Has had major psychiatric illness, which in the sponsor-investigator's opinion would compromise the participant's safety or compliance with the study procedures.
* Cannot communicate reliably with the sponsor-investigator or comply with study procedures.
* In the opinion of the sponsor-investigator, is unlikely to adhere to the requirements of the study or is unlikely to complete the full course of protocol required vaccination and observation.
* History of cancer malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or other malignancies with minimal risk of recurrence).
* History of acute polyneuropathy (e.g., Guillain-Barré syndrome)
* Chronic history of platelet count <75,000/µL.
* History of thrombosis with thrombocytopenia syndrome (TTS) or heparin-induced thrombocytopenia (HIS).
* History of capillary leak syndrome (CLS).
* Received pre-exposure prophylactic medications for COVID-19 that could interfere with assessments of any study-related endpoint
* History of myocarditis or pericarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Stegall, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park WD, Nair SS, Wadei HM, Liang Y, Smith BH, Abdelrheem A, Schinstock CA, Isham CR, Kumanovics A, Ahmad N, Simonson RB, Ryser MF, Tapia-Cealle G, Badley AD, Stegall MD. Responses of Kidney Transplant Recipients to Vaccination and Boosting. Mayo Clin Proc. 2025 Sep;100(9):1506-1518. doi: 10.1016/j.mayocp.2025.03.017. Epub 2025 Jul 16. PMID 40663029

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 468 subjects enrolled in the study; 49 were excluded as they didn't provide a screening serum sample. 29 subjects were excluded as they withdrew consent.
Groups:
- Initial Responders: Individuals who received the Pfizer or Moderna vaccines and had high levels of spike antibodies in their blood, received standard of care immunosuppressive (IS) medications.
- Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders: Individuals who had a spike protein test result less than 250 U/mL at the screening visit. Subjects received one dose of the Janssen Ad26.CoV2.S vaccine. After receiving the Janssen Ad26.CoV2.S vaccine, their spike protein test results were greater than or equal to 250 U/mL.
  Janssen Ad26.CoV2.S Vaccine: Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
- Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders: Individuals who had a spike protein test result less than 250 U/mL at the screening visit. Subjects received one dose of the Janssen Ad26.CoV2.S vaccine. After receiving the Janssen Ad26.CoV2.S vaccine, their spike protein test results were less than 250 U/mL. 28 days following the first dose of the Janssen Ad26.CoV2.S vaccine, subjects were given a second dose of Janssen Ad26.CoV2.S vaccine.
  Janssen Ad26.CoV2.S Vaccine: Single dose vaccine of 0.5 mL administered via intramuscular injection, typically in the deltoid muscle
Period: Initial Study Enrollment
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Started | 335 | 22 | 13 | 12 | 8
Completed | 335 | 22 | 13 | 12 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: First Janssen Vaccine Administration
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Started | 0 | 22 | 13 | 12 | 8
Completed | 0 | 22 | 13 | 12 | 8
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Janssen Vaccine Administration
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Started (12 participants met the criteria to receive the second dose of the Janssen Vaccine in the Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication arm, however 0 of those participants opted to receive the second dose of the vaccine.) | 0 | 0 | 13 | 0 | 0
Completed | 0 | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 8 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 8 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication | Total
Number analyzed (Participants) | 335 | 22 | 13 | 12 | 8 | 390
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (12.6) | 62.7 (11.2) | 61.5 (9.6) | 67.1 (6.9) | 63.4 (7.8) | 60.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 5 | 4 | 4 | 4 | 145
  Male | 207 | 17 | 9 | 8 | 4 | 245
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 3 | 1 | 0 | 1 | 34
  Not Hispanic or Latino | 306 | 18 | 11 | 12 | 6 | 353
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 0 | 1 | 0 | 0 | 7
  Asian | 9 | 0 | 0 | 0 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 0 | 0 | 0 | 3
  Black or African American | 29 | 0 | 1 | 2 | 1 | 33
  White | 279 | 22 | 10 | 10 | 5 | 326
  More than one race | 2 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 7 | 0 | 1 | 0 | 1 | 9
Region of Enrollment [Number; unit: participants]
  United States | 335 | 22 | 13 | 12 | 8 | 390

OUTCOME MEASURES:

1. Primary Outcome: Response to the Janssen Ad26.CoV2.S Vaccine in Subjects With Low Level Anti-COVID Spike Protein at Enrollment
Description: Number of patients with initial anti-COVID spike protein antibody levels >0 but <250U/ml at enrollment who receive the Janssen Ad26.CoV2.S vaccine who develop anti-COVID spike protein antibody levels greater than or equal to 250 U/mL at 28 days.
Time Frame: 28 days following first dose of Janssen Ad26.CoV2.S vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders
Number analyzed (Participants) | 22 | 13
Participants | 22 | 0

2. Primary Outcome: Response to the Janssen Ad26.CoV2.S Vaccine in Subjects With Undetectable Anti-COVID Spike Protein at Enrollment
Description: Number of patients with undetectable anti-COVID spike protein antibody level at enrollment who receive the Janssen Ad26.CoV2.S vaccine who develop anti-COVID spike protein antibody levels greater than or equal to 250 U/mL at 28 days.
Time Frame: 28 days following first dose of Janssen Ad26.CoV2.S vaccine
Measure: Count of Participants; unit: Participants
Arm/Group | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Number analyzed (Participants) | 12 | 8
Participants | 0 | 0

3. Secondary Outcome: Response to the Janssen Ad26.CoV2.S Vaccine in Subjects Who Had Low or Undetectable Levels of Anti-COVID Spike Protein After the First Dose of the Janssen Vaccine
Description: Number of subjects to achieve an anti-COVID spike protein antibody level greater than or equal to 250 U/mL 28 days after a second dose with the Janssen Ad26.CoV2.S vaccine.
Time Frame: 28 days after second dose of Janssen Ad26.CoV2.S vaccine, up to 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders
Number analyzed (Participants) | 5
Participants | 3

4. Secondary Outcome: Durability of Anti-COVID Spike Protein Antibody Levels in Patients Who Developed Any Level of Antibody Response After Receiving the Janssen Ad26.CoV2.S Vaccine.
Description: As measured by antibody levels from anti-COVID spike protein antibody tests.
Time Frame: 2 years
Population: No data was collected or analyzed on any subject for durability of anti-COVID spike protein antibody levels at 2 years as the study was terminated early.
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Incidence of COVID-19 Infection
Description: Number of subject infected with COVID-19 after enrollment. Criteria for suspected COVID includes: positive reverse transcription-polymerase chain reaction (RT-PCR) result for SARS-CoV-2 OR New onset or worsening of any one of the following symptoms, which lasts for at least 24 hours, not otherwise explained: headache, malaise, myalgia, chest congestion, cough, runny nose, shortness of breath or difficulty breathing (resting or on exertion), sore throat, wheezing, eye irritation or discharge, chills, fever (≥ 38.0°C or ≥ 100.4°F), pulse oximetry value ≤95% (which is a decrease from baseline), heart rate ≥90 bpm at rest (which is an increase from baseline), GI symptoms, neurologic symptoms, red or bruised looking toes, skin rash, taste loss or new/changing sense of smell, symptoms of blood clots, confusion, bluish lips or face, clinical suspicion or judgement by sponsor-investigator of symptoms suggestive for COVID-19.
Time Frame: 2 years
Population: No data was collected or analyzed on any subject for incidence of COVID-19 infection at 2 years as the study was terminated early.
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through study completion, approximately 2 months.
Description: This study defined an adverse event as any (S)AEs that are related to study procedures. Adverse events were collected through participant diaries and follow-up remote visits.
Arm/Group | Initial Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Responders | Low Levels (LL) Spike Antibodies: Janssen Vaccine Non-Responders | Undetectable Levels (UL) Spike Antibodies: Maintain Immunosuppression Medication | Undetectable Levels (UL) Spike Antibodies: Change Immunosuppression Medication
All-Cause Mortality (participants affected / at risk) | 0/335 | 0/22 | 0/13 | 0/12 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/335 | 0/22 | 0/13 | 0/12 | 0/8
Other Adverse Events (participants affected / at risk) | 0/335 | 0/22 | 0/13 | 0/12 | 0/8

LIMITATIONS AND CAVEATS:
This study was terminated early due to Janssen Biotech, Inc withdrawing the emergency use authorization from the FDA on May 22, 2023, as there was no demand for the new lots of Janssen COVID-19 vaccine in the United States. The vaccine was no longer being produced nor available by Janssen as of 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT05220397/Prot_SAP_000.pdf